CLINICAL TRIAL: NCT04154813
Title: Study on the Optimal Strategy of Chinese Patients With Bulimia Nervosa After Fluoxetine Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Huadong Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jue CHEN, Director of clinical psychology, Shanghai Mental Health Center
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BN001
Record Dates: First submitted 2019-10-28; First posted 2019-11-07 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Fluoxetine
MeSH Terms: interventions — Topiramate; Fluoxetine; Cognitive Behavioral Therapy; Dialectical Behavior Therapy

STUDY DESIGN:
Intervention Model Description: There is no evidence for patients who fail to respond to fluoxetine therapy to choose further treatment. As the result of fact, this study is proposed to adopt a two-stage sequential study design.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topiramate group (Experimental): If fluoxetine doesn't work after 3 months, randomly assigned to 3 groups, one group is topiramate group.During this group the initial dose of 25mg/day is rapidly increased to the target dose (100mg/day) or below the maximum tolerable dose if the patient can tolerate it.
  Interventions: Drug: Topiramate
- Fluoxetine+DBT group (Experimental): If fluoxetine doesn't work after 3 months, randomly assigned to 3 groups, one group is fluoxetine+DBT group. Group cognitive behavioral therapy was performed while fluoxetine was maintained. Target dose of fluoxetine is 60mg/day.Treatment was divided into three stages: the initial stage, the main stage and the end stage. The treatment was conducted once a week for a total of 12 times, followed by maintenance treatment for 6 months.
  Interventions: Drug: Fluoxetine; Behavioral: dialectical behavior therapy (DBT)
- Fluoxetine+CBT group (Experimental): If fluoxetine doesn't work after 3 months, randomly assigned to 3 groups, one group is fluoxetine+CBT group.Target dose of fluoxetine is 60mg/day. DBT therapy was performed while the original fluoxetine dose was maintained.The core treatment stage was 1 time per week, 12 times in total, and 6 months of maintenance treatment followed.
  Interventions: Drug: Fluoxetine; Behavioral: cognitive behavioral therapy (CBT)

INTERVENTIONS:
Drug: Topiramate — The initial dose of 25mg/d is rapidly increased to the target dose (100mg/d) or below the maximum tolerable dose if the patient can tolerate it.
  Arms: Topiramate group
Drug: Fluoxetine — Fluoxetine was increased from 20mg/d to the target dose (60mg/d) or below the maximum tolerable dose within 2 weeks.
  Arms: Fluoxetine+CBT group; Fluoxetine+DBT group
Behavioral: cognitive behavioral therapy (CBT) — CBT psychotherapy, once a week for three months.
  Arms: Fluoxetine+CBT group
Behavioral: dialectical behavior therapy (DBT) — DBT psychotherapy,once a week for three months.
  Arms: Fluoxetine+DBT group

SUMMARY:
Current treatment strategies for BN are limited. The total effective rate of pharmacotherapy and psychotherapy is only about 50%.The preliminary studies and clinical experience of this project indicate that :(1) fluoxetine, DBT and CBT were effective in controlling binge eating and purging behaviors in patients with BN;(2) the short-term efficacy of fluoxetine group is better than DBT group ;(3) treatment with fluoxetine is more convenient and easier to be accepted by Chinese patient and Chinese doctors. BN patients who had poor response to fluoxetine with adequate dosage and duration would receive a secondary treatment, and randomly assigned to three groups: topiramate, fluoxetine +CBT, fluoxetine +DBT.This study was designed as a multicenter randomized controlled study, in which 550 patients with bulimia were enrolled. During 1year of follow-up, the onset time, short-term and long-term efficacy, duration of treatment and the cost of each treatment strategies would be observed and compared.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) is a kind of chronic mental disorder which is easy to relapse, characterized by repeated binge eating, compensatory behaviors to prevent weight gain and excessive attention to one's own weight and body shape. Current treatment strategies for BN are limited. The total effective rate of pharmacotherapy and psychotherapy is only about 50%. All countries have listed SSRI drugs (fluoxetine 60mg/d has the most evidence from studies, and it is the only drug which has regulatory approval for the treatment of BN by FDA) and cognitive behavioral therapy (CBT) as the first-line treatment for BN. Other commonly used treatments include topiramate and dialectical behavior therapy (DBT).The preliminary studies and clinical experience of this project indicate that :(1) fluoxetine, DBT and CBT were effective in controlling binge eating and purging behaviors in patients with BN;(2) the short-term efficacy of fluoxetine group is better than DBT group ;(3) treatment with fluoxetine is more convenient and easier to be accepted by Chinese patient and Chinese doctors. Based on these factors above, this study was designed using fluoxetine as the initial treatment. However, there is no evidence for patients who fail to respond to fluoxetine therapy to choose further treatment. As the result of fact, this study is proposed to adopt a two-stage sequential study design.BN patients who had poor response to fluoxetine with adequate dosage and duration would receive a secondary treatment, and randomly assigned to three groups: topiramate, fluoxetine +CBT, fluoxetine +DBT.This study was designed as a multicenter randomized controlled study, in which 550 patients with bulimia were enrolled. During 1year of follow-up, the onset time, short-term and long-term efficacy, duration of treatment and the cost of each treatment strategies would be observed and compared. Based on the comprehensive evaluation of the advantages and disadvantage of each strategies, an evidence-based optimal strategy could be formed. The factors influencing the initial therapeutic effect and sequential therapeutic effect of BN would also be explored. If the expected results are obtained, it will provide strong support for the formulation of optimal clinical treatment strategy for BN.

ELIGIBILITY:
Inclusion Criteria:

* Have junior high school or above education level;
* Meet the diagnostic criteria of BN in DSM-5, body mass index (BMI)≥ 18.5kg /m2;
* Did not receive systematic nutrition treatment, psychiatric medication or any form of psychological treatment within 1 month before enrollment.
* Each patient must understand the nature of the study and sign an informed consent form.

Exclusion Criteria:

* those who meet DSM-5 except BN, such as substance abuse/dependence, depression, bipolar disorder, anxiety disorder, obsessive-compulsive disorder, high risk of suicide, strong destructive impulse or antisocial behavior;
* the patient has a serious primary or secondary physical disease, cognitive impairment, so that the patient can not complete the required symptom evaluation examination, psychological test;
* had received systematic nutritional treatment, individual and group psychotherapy;
* nearly 1 month to take neuroblockers, antidepressants, lithium, stimulants, antiepileptic drugs and other psychiatric drugs.
* for other reasons, the researchers considered it inappropriate to participate in this clinical trial.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 550 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination-Self-Report Questionnaire Version（EDE-Q） | Change from baseline the frequency of binge eating and clearing behaviors at 1 month, 2 months, 3 months, 6 months and 12 months.
  Has 41-item measure adapted from the Eating Disorder Examination (EDE), and four subscales of the EDE-Q: Restraint, Weight Concern, Shape Concern, and Eating Concern.

SECONDARY OUTCOMES:
Eating Disorder Inventory（EDI-II） | To evaluate the eating behavior and psychological changes of BN patients during treatment.1 month, 2 months, 3 months, 6 months, 12 months
  The EDI is a 64 item, self-report, multiscale measure designed for the assessment of psychological and behavioral traits common in eating disorder. The EDI consists of eight sub-scales measuring: 1) Drive for Thinness, 2) Bulimia, 3) Body Dissatisfaction, 4) Ineffectiveness, 5) Perfectionism, 6) Interpersonal Distrust, 7) Interoceptive Awareness and 8) Maturity Fears.
Beck Depression Inventory (BDI) | Evaluate the depression symptoms change from baseline at 1 month, 2 months, 3 months, 6 months and 12 months.
  use self-rating scale for depression, including 21 items of subjects such as emotional state, interests and hobbies, sleep quality, energy and spirit, and suicide risk.
Beck Anxiety Inventory (BAI) | Evaluate the anxiety symptoms change from baseline at 1 month, 2 months, 3 months, 6 months and 12 months.
  BAI has 21 self-assessment items, and subjects' degree of being bothered by various anxiety symptoms is taken as the assessment index, and the method of 4 grades is adopted.Its standard is "1" means none;"2" means mild, not much trouble;"3" means moderate, uncomfortable but tolerable;"4" means heavy, barely tolerable.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No